CLINICAL TRIAL: NCT01332318
Title: A Randomized, Double Blind, Active- and Placebo-Controlled, Parallel Group Safety Study Assessing Simulated Driving Performance in XP13512-(GSK1838262) Treated Patients With Restless Legs Syndrome
Brief Title: Simulated Driving Study in Restless Legs Syndrome
Acronym: XP083
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111463; XP083 (Other: XenoPort, Inc.)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2011-06

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): XP13512 Placebo + Diphenhydramine Placebo
  Interventions: Drug: Placebo
- XP13512 1200 mg (Experimental): XP13512 1200 mg/day + Diphenhydramine Placebo
  Interventions: Drug: XP13512
- XP13512 1800 mg (Experimental): XP13512 1800 mg/day + Diphenhydramine Placebo
  Interventions: Drug: XP13512
- Placebo + Diphenhydramine (Active Comparator): XP13512 Placebo + 50 mg Diphenhydramine
  Interventions: Drug: Diphenhydramine; Drug: Placebo

INTERVENTIONS:
Drug: XP13512 — XP13512 once daily for 16 days
  Other Names: GSK1838262; Gabapentin Enacarbil (GEn)
  Arms: XP13512 1200 mg; XP13512 1800 mg
Drug: Diphenhydramine — one 50 mg dose of diphenhydramine (DPH) on day 16
  Arms: Placebo + Diphenhydramine
Drug: Placebo — XP13512 placebo once daily for 16 days
  Arms: Placebo; Placebo + Diphenhydramine

SUMMARY:
This study was a multi center, randomized, double blind, active and placebo controlled, parallel group study to assess simulated driving performance in XP13512 treated subjects with Restless Legs Syndrome (RLS). Eligible subjects were randomized to receive a once daily dose of placebo (2 groups), XP13512 1200 mg, or XP13512 1800 mg for 16 days. On Day 16, one of the placebo groups also received one 50 mg dose of diphenhydramine (DPH) to assess the effects of an agent known to have sedative properties, while the other 3 groups received a DPH placebo.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, double blind, active and placebo controlled, parallel group study. Eligible subjects were randomized in a 1:1:1:1 ratio to 1 of the following 4 treatment groups:

A) XP13512 Placebo + Diphenhydramine Placebo (Pbo) B) XP13512 1200 mg/day + Diphenhydramine Placebo (1200 mg) C) XP13512 1800 mg/day + Diphenhydramine Placebo (1800 mg) D) XP13512 Placebo + 50 mg Diphenhydramine (Pbo/DPH)

ELIGIBILITY:
Inclusion Criteria:

* Men or women who were 21 through 65 years of age and fluent in English;
* Subjects with RLS, based on the IRLSSG Diagnostic Criteria;
* Currently a licensed and experienced driver who has driven an average of 3 or more times/week for the past 3 years;
* Able to successfully complete the 5 minute practice simulated driving test at Screening;
* History of RLS symptoms at least 15 nights in the prior month or, if on treatment, this frequency of symptoms before treatment was started;
* Total RLS severity score of 15 or greater on the IRLS Rating Scale;
* Documented RLS symptoms for at least 4 of the 7 consecutive evenings/nights Discontinuation of treatments for RLS (e.g., opioids, benzodiazepines, dopamine agonists and/or gabapentin) at least 2 weeks prior to Screening; -
* Body Mass Index of 34 or below;
* Estimated creatinine clearance of at least 60 mL/min;
* Agreed to maintain abstinence from alcohol and smoking throughout the entire study period;
* Agreed to maintain abstinence from caffeine from midnight of the day prior to and until the end of each Visit (Visits 2 to 4).

Exclusion Criteria:

* A sleep disorder (e.g., sleep apnea) other than RLS that may significantly affect the assessment of RLS;
* Current use of a sleeping medication or sedating medication;
* Current use of CNS stimulants;
* Neurologic disease or movement disorder;
* Other medical conditions which could affect RLS assessments;
* Significant medical history that may impair psychomotor coordination;
* Subjects who had clinically significant or unstable medical conditions;
* Serum ferritin level below 20 ng/mL;
* Subjects currently suffering from moderate or severe depression using the Diagnostic and Statistical Manual of Mental Disorders and Treatment IV (DSM IV TR);
* Subjects with a history of substance abuse (alcohol or drugs) or substance dependence within 12 months prior to enrollment;
* Shift workers or subjects who were not on normal day/night sleep cycles;
* Subjects who had smoked an average of greater than one half pack of cigarettes (or nicotine equivalent) per day within 30 days of the Screening Visit;
* Subjects who had consumed an average of >5 cups (i.e., 40 ounces) of caffeinated beverages per day within 20 days of the Screening Visit;
* Subjects with a history of allergy to gabapentin, diphenhydramine, or XP13512 excipients

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GEn Placebo and DPH Placebo: Oral gabapentin enacarbil (GEn) placebo taken once daily. Days 1 to 3: one placebo tablet. Days 4 to 7: two placebo tablets. Days 8 to 16: three placebo tablets. On Day 16, participants also took two capsules of diphenhydramine (DPH) placebo. On Day 17, participants entered a 7-day Taper Period. Days 17 to 20: two placebo tablets. Days 21 to 23: one placebo tablet.
- GEn 1200 mg and DPH Placebo: Oral GEn (XP13512/GSK1838262) 1200 milligrams (mg) taken once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 7: two ER tablets (600 mg GEn each). Days 8 to 16: two ER tablets (600 mg GEn each) and one placebo tablet. On Day 16, participants also took two capsules of DPH placebo. On Day 17, participants entered a 7-day Taper Period. Days 17 to 20: one ER tablet (600 mg GEn) and one placebo tablet. Days 21 to 23: one ER tablet (600 mg GEn).
- GEn 1800 mg and DPH Placebo: Oral GEn (XP13512/GSK1838262) 1800 mg taken once daily. Days 1 to 3: one ER tablet (600 mg GEn). Days 4 to 7: two ER tablets (600 mg GEn each). Days 8 to 16: three ER tablets (600 mg GEn each). On Day 16, participants also took two capsules of DPH placebo. On Day 17, participants entered a 7-day Taper Period. Days 17 to 20: two ER tablets (600 mg GEn each) and one placebo tablet. Days 21 to 23: one ER tablet (600 mg GEn).
- GEn Placebo and DPH 50 mg on Day 16: Oral GEn placebo taken once daily and oral DPH 50 mg taken once on Day 16. Days 1 to 3: one placebo tablet. Days 4 to 7: two placebo tablets. Days 8 to 16: three placebo tablets. On Day 16, participants also took two capsules of DPH (25 mg DPH each). On Day 17, participants entered a 7-day Taper Period. Days 17 to 20: two placebo tablets. Days 21 to 23: one placebo tablet.
Period: Overall Study
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Started | 34 | 32 | 34 | 30
Completed | 32 | 28 | 33 | 28
Not Completed | 2 | 4 | 1 | 2
Not completed — Adverse Event | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: There was one randomized participant (in the GEn 1200 mg and DPH Placebo group) who did not meet the criteria for inclusion in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16 | Total
Number analyzed (Participants) | 34 | 31 | 34 | 30 | 129
Age Continuous [Mean (Standard Deviation); unit: Years] — The Safety Population (all participants who received at least one dose [or a portion of a dose] of study drug) was used for all baseline characteristics. There was one randomized participant (in the GEn 1200 mg and DPH Placebo group) who did not meet the criteria for inclusion in the Safety Population.
  Years | 49.6 (11.40) | 46.8 (11.31) | 49.3 (10.27) | 40.6 (11.80) | 46.8 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population (all participants who received at least one dose [or any portion of a dose] of study drug) was used for all baseline characteristics. There was one randomized participant (in the GEn 1200 mg and DPH Placebo group) who did not meet the criteria for inclusion in the Safety Population.
  Participants
    Female | 20 | 21 | 17 | 19 | 77
    Male | 14 | 10 | 17 | 11 | 52
Race/Ethnicity, Customized [Number; unit: participants] — The Safety Population (all participants who received at least one dose [or any portion of a dose] of study drug) was used for all baseline characteristics. There was one randomized participant (in the GEn 1200 mg and DPH Placebo group) who did not meet the criteria for inclusion in the Safety Population.
  participants
    White or Caucasian | 34 | 31 | 33 | 30 | 128
    Other, Unknown | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day -1) in Overall Lane Position Variability (LPV) on Day 16 (Tmax)
Description: Lane position variability (LPV) was defined as the standard deviation of lane position, and was measured from the center line of the 26 foot wide 2-lane paved road to the center of the vehicle. Change from baseline in overall LPV was calculated as the Day 16 mean LPV over the 1-hour drive minus the Baseline mean LPV over the 1-hour drive. The Day 16 measurement is at the time of maximum concentration (Tmax) for both GEn and DPH.
Time Frame: Baseline (Day -1) and Day 16
Population: Modified Intent-to-Treat (MITT) Population: all participants in the Safety Population who completed at least one Baseline and one End of Study (Days 14-16) simulated driving assessment. The number of participants assessed at each study day varies due to incomplete/missing data.
Measure: Least Squares Mean (Standard Error); unit: feet
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 30 | 28 | 33 | 28
feet | -0.10 (0.06) | 0.15 (0.06) | 0.15 (0.06) | 0.16 (0.06)
Statistical Analysis 1: Comparison: GEn Placebo and DPH Placebo vs GEn 1200 mg and DPH Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 0.15, 95% CI [0.08 to 0.42], Standard Error of Mean 0.06 — An Analysis of Covariance (ANCOVA) model, including terms for treatment, pooled study site, visit, and treatment by visit interaction, was used to calculate the adjusted mean difference and confidence interval. Arm 2 minus Arm 1
Statistical Analysis 2: Comparison: GEn Placebo and DPH Placebo vs GEn 1800 mg and DPH Placebo; Test type: Superiority or Other; Least Squares Mean Difference = 0.15, 95% CI [0.09 to 0.41], Standard Error of Mean 0.06 — An Analysis of Covariance (ANCOVA) model, including terms for treatment, pooled study site, visit, and treatment by visit interaction, was used to calculate the adjusted mean difference and confidence interval. Arm 3 minus Arm 1
Statistical Analysis 3: Comparison: GEn Placebo and DPH Placebo vs GEn Placebo and DPH 50 mg on Day 16; Test type: Superiority or Other; Least Squares Mean Difference = 0.16, 95% CI [0.09 to 0.42], Standard Error of Mean 0.06 — An Analysis of Covariance (ANCOVA) model, including terms for treatment, pooled study site, visit, and treatment by visit interaction, was used to calculate the adjusted mean difference and confidence interval. Arm 4 minus Arm 1

2. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in Overall Lane Position Variability (LPV)
Description: Lane position variability (LPV) was defined as the standard deviation of lane position, and was measured from the center line of the 26 foot wide 2-lane paved road to the center of the vehicle. Change from baseline in overall LPV was calculated as the Day 14 (in the evening) or Day 15 (in the morning after GEn dosed at 5 PM) mean LPV over the 1-hour drive minus the Baseline (Day -1 or Day 1) mean LPV over the 1-hour drive.
Time Frame: Baseline (Days -1 and 1) and Days 14 and 15
Population: Modified Intent-to-Treat (MITT) Population. The number of participants assessed at each study day varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
feet
  Day 14, n=33, 28, 33, 28 | -0.06 (0.17) | 0.17 (0.43) | -0.01 (0.28) | -0.08 (0.15)
  Day 15, n=32, 28, 31, 27 | -0.01 (0.14) | 0.13 (0.40) | 0.02 (0.32) | -0.10 (0.19)

3. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in Overall Average Lane Position
Description: Lane position was measured from the center line of the 26 foot wide 2-lane paved road to the center of the vehicle. Change from baseline in overall average lane position was calculated as the Day 14 (in the evening), 15 (in the morning after GEn dosed at 5 PM), or 16 (assessment at Tmax of GEn and DPH) mean lane position over the 1-hour drive minus the Baseline (Days -1 and 1) mean lane position over the 1-hour drive.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
feet
  Day 14, n=33, 28, 33, 28 | 0.05 (0.35) | -0.02 (0.64) | 0.03 (0.32) | 0.08 (0.29)
  Day 15, n=32, 28, 31, 27 | 0.01 (0.35) | 0.12 (0.39) | 0.04 (0.34) | 0.04 (0.28)
  Day 16, n=30, 28, 33, 28 | 0.17 (0.44) | 0.13 (0.48) | 0.14 (0.32) | 0.08 (0.31)

4. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in Overall Speed Variability
Description: Speed variability was defined as the standard deviation of the speed (measured in miles per hour). Participants were instructed to maintain a speed of 55 miles per hour during the test drive. Change from baseline in overall speed variability was calculated as the Day 14 (in the evening), 15 (in the morning), or 16 (at Tmax of GEn and DPH) mean speed variability over the 1-hour drive minus the Baseline (Days -1 and 1) mean speed variability over the 1-hour drive.
Time Frame: Baseline (Day -1) and Days 14 and 16; baseline (Day 1) and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: miles per hour
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
miles per hour
  Day 14, n=33, 28, 33, 28 | -0.22 (0.63) | -0.19 (1.42) | -0.32 (1.17) | -0.47 (0.96)
  Day 15, n=32, 28, 31, 27 | -0.26 (0.48) | 0.43 (2.22) | -0.07 (0.69) | -0.33 (0.43)
  Day 16, n=30, 28, 33, 28 | -0.54 (0.55) | -0.12 (2.02) | 0.23 (1.95) | -0.08 (1.11)

5. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in Overall Average Speed
Description: Participants were instructed to maintain a speed of 55 miles per hour during the driving assessment. Change from baseline in overall average speed was calculated as the Day 14 (in the evening), 15 (in the morning), or 16 (at Tmax of GEn and DPH) mean speed over the 1-hour drive minus the Baseline (Days -1 and 1) mean speed over the 1-hour drive.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: miles per hour
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
miles per hour
  Day 14, n=33, 28, 33, 28 | 1.24 (1.49) | 0.66 (1.34) | 0.42 (1.43) | 0.12 (1.51)
  Day 15, n=32, 28, 31, 27 | 0.75 (1.75) | 0.33 (0.97) | 0.30 (1.12) | 0.37 (1.04)
  Day 16, n=30, 28, 33, 28 | 1.70 (1.92) | 0.90 (1.58) | 0.92 (1.64) | 0.84 (1.64)

6. Secondary Outcome: Number of Participants With the Indicated Number of Simulated Crashes on Days 14 (Evening), 15 (Morning After Dose), and 16 (Tmax)
Description: A simulated crash was defined as a collision with an oncoming car or obstacle (e.g., tree) or when the distance to the center line was greater than 18 feet on either side of the road.
Time Frame: Days 14, 15, and 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
participants
  Day 14; 1 Crash, n=33, 28, 33, 28 | 2 | 1 | 0 | 1
  Day 14; 2 Crashes, n=33, 28, 33, 28 | 2 | 2 | 0 | 0
  Day 14; 3 Crashes, n=33, 28, 33, 28 | 0 | 0 | 1 | 0
  Day 14; 4 Crashes, n=33, 28, 33, 28 | 0 | 1 | 0 | 0
  Day 14; 5 Crashes, n=33, 28, 33, 28 | 0 | 1 | 0 | 0
  Day 14; 13 Crashes, n=33, 28, 33, 28 | 0 | 1 | 0 | 0
  Day 15; 1 Crash, n=33, 28, 31, 28 | 1 | 4 | 1 | 0
  Day 15; 2 Crashes, n=33, 28, 31, 28 | 0 | 3 | 0 | 0
  Day 15; 4 Crashes, n=33, 28, 31, 28 | 0 | 2 | 0 | 0
  Day 15; 13 Crashes, n=33, 28, 31, 28 | 0 | 1 | 0 | 0
  Day 16; 1 Crash, n=30, 28, 33, 28 | 0 | 5 | 3 | 2
  Day 16; 3 Crashes, n=30, 28, 33, 28 | 0 | 1 | 2 | 0
  Day 16; 4 Crashes, n=30, 28, 33, 28 | 0 | 1 | 0 | 0
  Day 16; 5 Crashes, n=30, 28, 33, 28 | 0 | 0 | 0 | 1
  Day 16; 13 Crashes, n=30, 28, 33, 28 | 0 | 0 | 1 | 0
  Day 16; 17 Crashes, n=30, 28, 33, 28 | 0 | 1 | 0 | 0

7. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in Brake Reaction Time
Description: Brake reaction time was assessed as the time it took for each participant to move their foot off the accelerator and onto the brake pedal after the appearance of a stop sign on the simulation screen. Change from baseline was calculated as the Day 14, 15, or 16 mean reaction time minus the Baseline (Days -1 and 1) mean reaction time.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 27
seconds
  Day 14, n=33, 25, 32, 27 | -0.04 (0.08) | -0.07 (0.09) | -0.03 (0.12) | -0.04 (0.12)
  Day 15, n=32, 25, 30, 25 | -0.00 (0.07) | -0.03 (0.08) | -0.01 (0.15) | -0.05 (0.10)
  Day 16, n=30, 28, 33, 27 | -0.04 (0.10) | -0.05 (0.15) | -0.03 (0.10) | -0.03 (0.16)

8. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in the Alertness Visual Analog Scale (VAS) Score
Description: Alertness VAS was completed immediately before and after each simulated driving assessment. Participants indicated their alertness by marking a vertical line on a horizontal scale anchored by responses "extremely sleepy" and "extremely alert." VAS score was determined by measuring the distance in millimeters (mm) from the left hand end of the line to the point the participant marked. Scores ranged from 0-100 mm, with higher scores indicating more alertness and lower scores indicating more sleepiness. Change score was calculated as the Day 14, 15, or 16 VAS score minus the Baseline VAS score.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: Modified Intent-to-Treat (MITT) Population. Varying numbers of participants did not complete either the pre- or post-drive VAS at either Baseline or the day of assessment; as such, the number of participants analyzed varies by day.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
millimeters
  Day 14; Pre-Drive, n=33, 28, 32, 28 | 4.5 (22.98) | -2.6 (25.43) | -3.5 (29.39) | -3.1 (20.99)
  Day 14; Post-Drive, n=33, 28, 32, 28 | 7.7 (21.72) | 3.2 (21.76) | 3.3 (21.48) | -3.0 (22.62)
  Day 14; Post-Pre Drive Difference, n=33,28,32,28 | 3.1 (26.04) | 5.9 (20.69) | 4.9 (25.09) | 0.1 (24.66)
  Day 15; Pre-Drive, n=33, 27, 33, 28 | 1.5 (15.56) | 0.2 (26.98) | 7.2 (21.53) | 0.4 (22.10)
  Day 15; Post-Drive, n=33, 27, 32, 27 | -3.2 (18.92) | -6.1 (28.44) | 4.8 (21.08) | -3.1 (22.97)
  Day 15; Post-Pre Drive Difference, n=33,27,32,27 | -4.7 (22.22) | -6.3 (24.55) | -2.2 (27.45) | -3.7 (33.84)
  Day 16; Pre-Drive, n=32, 28, 33, 28 | 6.3 (23.44) | 0.8 (32.79) | -8.8 (27.61) | -11.8 (24.00)
  Day 16; Post-Drive, n=31, 28, 33, 28 | 14.3 (22.23) | -3.6 (32.01) | -7.5 (26.17) | -14.0 (29.25)
  Day 16; Post-Pre Drive Difference, n=31,28,33,28 | 7.7 (22.38) | -4.5 (36.14) | 1.3 (34.13) | -2.3 (23.91)

9. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) in the Epworth Sleepiness Scale (ESS) Total Score
Description: The Epworth Sleepiness Scale (ESS) is a questionnaire designed to evaluate daytime sleepiness. Participants were asked to rate how likely they were to doze or fall asleep during 8 activities on a scale of 0 ("would never do") to 3 ("high chance of dozing"). The total score ranges from 0-24, with a score greater than 10 representing excessive daytime sleepiness (an increased chance of dozing). Change from baseline was calculated as the Day 14 total score minus the Baseline total score.
Time Frame: Baseline (Day -1) and Day 14
Population: Modified Intent-to-Treat (MITT) Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale | -2.6 (3.22) | -2.3 (5.61) | -2.4 (5.04) | -2.4 (4.88)

10. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Composite Score
Description: The BAC was designed as a comprehensive measure of cognitive function, including 6 individual tests: Verbal Memory Recall, Digit Sequencing, Token Motor Task, Verbal Fluency, Symbol Coding, and Tower of London. The composite/total BAC score is calculated by scoring each individual test, comparing each score to a healthy control sample (matched for sex and age category) to create z-scores, summing the z-scores, and rescaling the sum. The composite score range is -2127.8 to 1878.8, with higher scores indicating better cognition.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 4.6 (5.64) | 5.3 (7.01) | 5.3 (6.88) | 7.0 (6.25)
  Day 15, n=33, 28, 33, 28 | 4.8 (5.39) | 3.4 (4.59) | 0.2 (6.61) | 4.8 (4.66)
  Day 16, n=32, 28, 33, 28 | 7.2 (7.24) | 9.1 (8.98) | 7.1 (8.34) | 10.7 (6.05)

11. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Verbal Memory Test Score
Description: Participants were presented with 15 words and asked to recall as many as possible; the procedure was repeated 5 times. The total number of words recalled correctly across the 5 administrations of the list was the participant's Verbal Memory Recall score (range: 0-75). The scaled test score was calculated as ((BAC component raw test score - healthy control sample test mean)/healthy control sample test standard deviation); a healthy control sample was matched to the participant's sex and age category. The scaled test score range is -7.37 to 4.86; higher scaled scores indicate better cognition.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.1 (0.77) | 0.1 (0.83) | 0.2 (0.82) | 0.1 (0.94)
  Day 15, n=33, 28, 33, 28 | 0.2 (0.63) | 0.1 (0.75) | -0.0 (0.93) | 0.1 (0.80)
  Day 16, n=32, 28, 33, 28 | -0.2 (0.78) | -0.1 (0.88) | 0.1 (0.97) | 0.0 (0.92)

12. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Digit Sequencing Score (DSS)
Description: Participants (par.) were presented with sets of numbers of increasing length and asked to tell the experimenter the numbers in order from lowest to highest. The task has 7 levels; the first level had 2 digits in the set (e.g., 5, 2); the second level had 3 digits in the set, etc. The number of times the par. correctly arranged the numbers was recorded as the score for each level. The DSS is the sum of the 7 level scores (range: 0-28). The scaled test score was calculated as indicated for the Verbal Memory Test and ranges from -6.68 to 2.73; higher scaled scores indicate better cognition.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.3 (0.84) | 0.2 (0.90) | 0.4 (0.75) | 0.3 (0.80)
  Day 15, n=33, 28, 33, 28 | 0.2 (0.83) | 0.3 (0.86) | -0.2 (0.72) | 0.1 (0.69)
  Day 16, n=32, 28, 33, 28 | 0.3 (0.79) | 0.4 (0.66) | 0.5 (0.73) | 0.7 (0.75)

13. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Token Motor Task Test Score
Description: Participants were given 100 plastic tokens and asked to place them in a container, 2 at a time, as quickly as possible for 60 seconds. The number of tokens correctly placed in the container was the Token Motor Task score (range: 0-100). The BAC was conducted prior to each simulated driving test. The Token Motor Task scaled test score was calculated as indicated for the Verbal Memory Test. Change from baseline was calculated as the Day composite score minus the Baseline composite score. The scaled test score range is -6.95 to 3.35, with higher scaled scores indicating better cognition.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.2 (1.03) | 0.4 (1.06) | 0.2 (1.29) | 0.3 (0.89)
  Day 15, n=33, 28, 33, 28 | 0.4 (1.12) | -0.0 (0.93) | -0.2 (0.86) | 0.2 (0.67)
  Day 16, n=32, 28, 33, 28 | 0.4 (1.08) | 0.4 (1.04) | 0.1 (1.34) | 0.4 (1.09)

14. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Verbal Fluency Test Score
Description: Verbal Fluency included one semantic fluency and two letter fluency tasks. Participants were given 60 seconds to name as many words as possible within a given semantic category (supermarket items), and in two separate trials, participants were given 60 seconds to generate as many words as possible that began with a given letter. The total number of words from all of the 3 trials was the Verbal Fluency score (range: 0-150). The scaled test score was calculated as indicated for the Verbal Memory Test. The scaled test score range is -5 to 10.83; higher scaled scores indicate better cognition.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.2 (0.91) | 0.5 (0.84) | 0.4 (0.76) | 0.6 (0.68)
  Day 15, n=33, 28, 33, 28 | 0.4 (0.65) | 0.1 (0.65) | 0.2 (0.68) | 0.4 (0.87)
  Day 16, n=32, 28, 33, 28 | 0.7 (1.04) | 0.7 (0.83) | 0.4 (0.97) | 0.9 (0.98)

15. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Symbol Coding Test Score
Description: Participants were given a list of numbers (numerals 1-9) that were each associated with a unique symbol. Participants decoded a list of 110 symbols as quickly as possible in 90 seconds. The total number of symbols correctly decoded was the Symbol Coding Score (range: 0-110). The Symbol Coding scaled test score was calculated as indicated for the Verbal Memory Test. Change from baseline was calculated as the Day composite score minus the Baseline composite score. The scaled test score range is -7 to 10.08, with higher scaled scores indicating better cognition.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.6 (0.57) | 0.6 (0.87) | 0.5 (0.72) | 0.6 (0.85)
  Day 15, n=33, 28, 33, 28 | 0.5 (0.85) | 0.5 (0.78) | -0.0 (1.04) | 0.4 (0.78)
  Day 16, n=32, 28, 33, 28 | 1.3 (0.92) | 1.4 (1.28) | 1.0 (0.95) | 1.3 (0.81)

16. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Brief Assessment of Cognition (BAC) Scaled Tower of London (TOL) Score
Description: Participants (par.) were asked to look at 2 pictures simultaneously; each picture showed 3 different colored balls arranged on 3 pegs. Par. were to estimate the number of times the balls in 1 picture would have to be moved to make the arrangement of balls identical to that of the second picture. Par. were allowed 20 seconds to respond to each pair of pictures. The number of correct items was the TOL Score (range: 0-22). The TOL scaled test score was calculated as indicated for the Verbal Memory Test. The scaled test score range is -7.53 to 2.76; higher scaled scores indicate better cognition.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Number analyzed (Participants) | 33 | 28 | 33 | 28
scores on a scale
  Day 14, n=33, 28, 33, 28 | 0.3 (0.59) | 0.2 (1.03) | 0.3 (1.17) | 0.5 (0.95)
  Day 15, n=33, 28, 33, 28 | 0.2 (0.65) | 0.3 (0.90) | 0.4 (0.89) | 0.5 (1.30)
  Day 16, n=32, 28, 33, 28 | 0.1 (0.73) | 0.5 (0.91) | 0.5 (0.96) | 0.6 (0.92)

17. Secondary Outcome: Mean Change From Baseline (Day -1) at Day 14 in the International Restless Legs Syndrome (IRLS) Rating Scale Total Score
Description: The IRLS Rating scale is a measure of RLS disease severity and reflects the participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Items are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total score ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement.
Time Frame: Baseline (Day -1) and Day 14
Population: Modified Intent-to-Treat (MITT) Population. Participants in the "GEn placebo and DPH placebo" and the "GEn placebo and DPH 50 mg on Day 16" arms have been combined into the "GEn placebo and DPH" group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- GEn Placebo and DPH: The GEn placebo and DPH placebo participants were pooled with the GEn placebo and DPH 50 mg on Day 16 participants. Days 1 to 3: one placebo tablet. Days 4 to 7: two placebo tablets. Days 8 to 16: three placebo tablets. On Day 16, participants either took two capsules of DPH placebo or two capsules DPH (25 mg DPH each). On Day 17, participants entered a 7-day Taper Period. Days 17 to 20: two placebo tablets. Days 21 to 23: one placebo tablet.
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
scores on a scale | -7.6 (7.63) | -12.4 (9.93) | -13.1 (8.09)

18. Secondary Outcome: Number of Participants in Each Category of the Investigator-Rated Clinician Global Impression of Improvement (CGI-I) Scale at Day 14
Description: The CGI scale is a widely used tool designed to allow clinicians to rate the severity of illness and the change of the disease severity over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline.
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants
  Very Much Improved, score of 1 | 7 | 10 | 15
  Much Improved, score of 2 | 15 | 7 | 8
  Minimally Improved, score of 3 | 19 | 7 | 6
  No Change, score of 4 | 15 | 4 | 4
  Minimally Worse, score of 5 | 4 | 0 | 0
  Much Worse, score of 6 | 1 | 0 | 0
  Very Much Worse, score of 7 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants Who Responded to Treatment Based on Scores on the Investigator-Rated CGI-I at Day 14
Description: The investigator-rated CGI-I is a clinician-rated assessment designed to allow clinicians to rate the change of their participant's disease severity over time based on a seven-point scale, with a score of 1 being "very much improved," and a score of 7 being "very much worse" compared to baseline. For this endpoint, "response" was defined as a rating of "very much improved" or "much improved" (score of 1 or 2 on the scale) compared to baseline.
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants | 22 | 17 | 23

20. Secondary Outcome: Number of Participants in Each Category of the Participant-Rated Clinician Global Impression of Improvement (CGI-I) Scale at Day 14
Description: The participant-rated CGI-I scale is a self-rated assessment designed to allow participants to rate the change of their disease severity over time based on a seven-point scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse".
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants
  Very Much Improved, score of 1 | 7 | 9 | 14
  Much Improved, score of 2 | 16 | 11 | 9
  Minimally Improved, score of 3 | 14 | 3 | 6
  No Change, score of 4 | 17 | 3 | 4
  Minimally Worse, score of 5 | 5 | 2 | 0
  Much Worse, score of 6 | 2 | 0 | 0
  Very Much Worse, score of 7 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants Who Responded to Treatment Based on Scores on the Participant-Rated CGI-I at Day 14
Description: The participant-rated CGI-I is a self-rated assessment designed to allow participants to rate the change of their disease severity over time based on a seven-point scale, with a score of 1 being "very much improved," and a score of 7 being "very much worse." "Response" was defined as a rating of "very much improved" or "much improved" (score of 1 or 2 on the scale).
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants | 23 | 20 | 23

22. Secondary Outcome: Median Time to Onset of a Participant's First RLS Symptoms Using the 24-hour RLS Symptom Record at Day 14
Description: The 24-Hour RLS Record is a diary in which participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-min increments beginning at 8AM on the day prior to the visit. For Arms 2 and 3, upper limits of the confidence intervals are not available, as they are beyond the 24-hour time frame.
Time Frame: Day 14
Population: Modified Intent-to-Treat (MITT) Population. Participants in the
Measure: Median (95% Confidence Interval); unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants | 7.0 [3.5 to 13.0] | 14.3 [7.5 to NA] — The upper limit of the confidence interval is not available, as it is beyond the 24-hour time frame. | 15.5 [13.5 to NA] — The upper limit of the confidence interval is not available, as it is beyond the 24-hour time frame.

23. Secondary Outcome: Percentage of Participants With no Reported RLS Symptoms During the 24-hour RLS Record at Day 14
Description: The 24-Hour RLS Record is a diary in which participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-min increments beginning at 8AM on the day prior to the visit.
Time Frame: Day 14
Population: Modified Intent-to-Treat (MITT) Population. Participants in the
Measure: Number; unit: percentage of participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
percentage of participants | 9.84 | 35.71 | 42.42

24. Secondary Outcome: Number of Participants With no Reported RLS Symptoms During Each of the 4-hour Periods From the 24-hour RLS Record at Day 14
Description: The 24-Hour RLS Record is a diary in which participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-minute increments. The period was divided into 7 four-hour intervals (8 AM to 12 PM, 12 PM to 4 PM, 4 PM to 8 PM, 6 PM to 10 PM, 8 PM to 12 Midnight, Midnight to 4 AM, and 4 AM to 8 AM).
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants
  8 AM to 12 PM | 37 | 21 | 27
  12 PM to 4 PM | 35 | 20 | 23
  4 PM to 8 PM | 36 | 19 | 26
  6 PM to 10 PM | 27 | 18 | 23
  8 PM to 12 AM | 18 | 13 | 18
  12 AM to 4 AM | 24 | 17 | 24
  4 AM to 8 AM | 39 | 23 | 26

25. Secondary Outcome: Number of Participants With the Indicated Post Sleep Questionnaire (PSQ) Responses at Day 14
Description: The PSQ is designed to evaluate sleep quality, ability to function, and the degree to which RLS symptoms interfere with sleep.
Time Frame: Day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
participants
  Sleep Quality: Excellent | 9 | 5 | 14
  Sleep Quality: Reasonable | 31 | 18 | 17
  Sleep Quality: Poor | 21 | 5 | 2
  Ability to Function: Excellent | 8 | 6 | 11
  Ability to Function: Good | 32 | 17 | 18
  Ability to Function: Moderate | 20 | 5 | 4
  Ability to Function: Poor | 1 | 0 | 0
  0 Nights with RLS Symptoms | 8 | 8 | 10
  1-2 Nights with RLS Symptoms | 12 | 7 | 9
  3-4 Nights with RLS Symptoms | 17 | 6 | 8
  5-6 Nights with RLS Symptoms | 13 | 1 | 3
  7 Nights with RLS Symptoms | 11 | 6 | 3
  0 Awakenings/Night due to RLS | 10 | 7 | 8
  1-2 Wakenings/Night due to RLS | 41 | 18 | 23
  3-4 Awakenings/Night due to RLS | 8 | 2 | 1
  5+ Awakenings/Night due to RLS | 2 | 1 | 1
  0 Hours Awake/Night due to RLS | 53 | 23 | 31
  <1 Hour Awake/Night due to RLS | 3 | 4 | 0
  1-<2 Hours Awake/Night due to RLS | 3 | 0 | 0
  2-<3 Hours Awake/Night due to RLS | 2 | 1 | 2
  3+ Hours Awake/Night due to RLS | 0 | 0 | 0

26. Secondary Outcome: Mean Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) on the Pittsburgh Sleep Diary (PghSD) Sleep Onset Items
Description: The PghSD assessed participant's previous night's sleep. Change from baseline was calculated as the Day 14 (in the evening), 15 (in the morning), and 16 (at Tmax of GEn and DPH) value minus the Baseline (Days -1 and 1) value. Latency to sleep onset (time to fall asleep) and wake time after sleep onset are expressed in minutes.
Time Frame: Baseline (Days -1and 1) and Days 14, 15, and 16
Population: Modified Intent-to-Treat (MITT) Population. Participants in the "GEn placebo and DPH placebo" and the "GEn placebo and DPH 50 mg on Day 16" arms have been combined into the "GEn placebo and DPH" group. The number of participants assessed for each PghSD question at each study day varies due to incomplete/missing data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
minutes
  Day 14; Latency to Sleep Onset, n=61, 28, 33 | -8.1 (54.74) | -3.2 (62.96) | -25.7 (60.32)
  Day 14; Wake Time After Sleep Onset, n=59, 26, 33 | -14.0 (45.46) | -23.3 (41.11) | -26.9 (45.18)
  Day 15; Latency to Sleep Onset n=61, 28, 33 | -8.7 (57.28) | -14.9 (54.05) | -35.8 (59.02)
  Day 15; Wake Time After Sleep Onset, n=60, 28, 33 | 4.9 (61.11) | -30.8 (51.97) | -14.8 (64.07)
  Day 16; Latency to Sleep Onset, n=60, 28, 23 | -17.3 (46.6) | -3.3 (55.67) | -19.3 (52.76)
  Day 16; Wake Time After Sleep Onset, n=59, 26, 33 | -15.8 (55.44) | -26.3 (29.50) | -9.9 (60.58)

27. Secondary Outcome: Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in the Pittsburgh Sleep Diary (PghSD) Total Sleep Time Item
Description: The PghSD assessed a participant's previous night's sleep. Change from baseline was calculated as the Day 14 (in the evening), 15 (in the morning after dose), and 16 (at Tmax)value minus the Baseline (Days -1 and 1) value. Total sleep time is expressed in hours.
Time Frame: Baseline (Days -1 and 1) and Days 14, 15, and 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
hours
  Day 14, n=59, 26, 33 | 0.3 (1.60) | 0.2 (1.82) | 1.0 (2.39)
  Day 15, n=60, 28, 33 | -0.2 (2.10) | 0.2 (1.24) | 0.3 (1.54)
  Day 16, n=59, 26, 33 | 0.5 (1.82) | 0.3 (1.32) | 0.4 (1.91)

28. Secondary Outcome: Mean Change From Baseline (Day -1) to Day 14 (Evening) and Day 16 (at Tmax) and Change From Baseline (Day 1) to Day 15 (Morning After Dose) in the Pittsburgh Sleep Diary (PghSD) Sleep Quality
Description: The PghSD assessed a participant's previous night's sleep. Sleep quality was assessed using a Visual Analogue Scale (VAS). Participants indicated their sleep quality by marking a vertical line on a horizontal scale anchored by responses "very bad" and "very good." VAS score was determined by measuring the distance in millimeters (mm) from the left hand end of the line to the point that the participant marked. Scores ranged from 0 to 100 mm with higher scores indicating better sleep quality and lower scores indicating worse sleep quality.
Time Frame: Baseline (Day -1and 1) and Days 14, 15, and 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | GEn Placebo and DPH | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo
Number analyzed (Participants) | 61 | 28 | 33
millimeters
  Day 14, n=61, 28, 33 | 21.2 (29.47) | 29.9 (30.76) | 35.1 (28.84)
  Day 15, n=61, 28, 33 | 11.8 (27.30) | 24.6 (29.15) | 18.0 (24.82)
  Day 16, n=59, 28, 33 | 20.7 (25.01) | 27.4 (24.11) | 16.7 (28.86)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs): First dose of randomized study medication through end of Taper Phase (Day 23). Any Serious Adverse Event (SAE) reported up to 30 days after last dose was also reported.
Description: TEAEs were AEs reported in the Safety Population from the time the first dose of study drug was administered to the end of the Taper Phase (Day 23). AEs were considered TEAEs if the onset date or a reported change in severity (for ongoing events) occurred after Randomization.
Arm/Group | GEn Placebo and DPH Placebo | GEn 1200 mg and DPH Placebo | GEn 1800 mg and DPH Placebo | GEn Placebo and DPH 50 mg on Day 16
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 10/34 | 16/31 | 21/34 | 11/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GEn Placebo and DPH Placebo (N=34) | GEn 1200 mg and DPH Placebo (N=31) | GEn 1800 mg and DPH Placebo (N=34) | GEn Placebo and DPH 50 mg on Day 16 (N=30)
Somnolence (Nervous system disorders) | 1 | 8 | 13 | 2
Headache (Nervous system disorders) | 3 | 5 | 4 | 4
Dizziness (Nervous system disorders) | 3 | 4 | 4 | 2
Fatigue (General disorders) | 1 | 2 | 4 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Balance Disorder (Nervous system disorders) | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Motion Sickness (Ear and labyrinth disorders) | 1 | 0 | 2 | 0
Restless Legs Syndrome (Nervous system disorders) | 3 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Feeling Abnormal (General disorders) | 0 | 0 | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.